CLINICAL TRIAL: NCT01778179
Title: Safety and Efficacy of a Triple Combination Cream as Adjuvant Treatment of Solar Lentigines With Cryotherapy.
Brief Title: A Fixed Triple Combination Cream for Solar Lentigines Associated to Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-03
Record Dates: First submitted 2013-01-04; First posted 2013-01-29 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Solar Lentigines
Keywords: Lentigines; Cryotherapy; hyperpigmentation
MeSH Terms: conditions — Lentigo; Hyperpigmentation | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Subjects (group 1) will be treated daily for their solar lentigines with the investigational drug (Tri-Luma® cream) plus sunscreen for 2 weeks. At week 2, all the subjects will have the solar lentigines treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (From Week 2 up to Week 13)
  * Topical antibiotic treatment phase (Week 2 up to Week 5 - visit 2 to visit 3): At week 2, all the subjects will start to apply a topical antibiotic (Neomycin/Nebacetin® ointment) for the next 3 weeks.
  * Treatment phase 2 (from week 5 up to week 13 - visit 3 up to visit 5):
  The investigational drug (Tri-Luma® cream) plus sunscreen will be applied again (group 1) for a minimum of 4 weeks and up to 8 weeks, according to the Global Improvement of solar lentigines and absence of PIH.
  Interventions: Drug: Tri-luma; Procedure: Cryotherapy (CRY-AC3® device)
- Group 2 (Placebo Comparator): Subjects (group 2) will be treated daily for their solar lentigines with sunscreen alone for 2 weeks. At week 2, all the subjects will have the solar lentigines will treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (Week 2 up to Week 13)
  * Topical antibiotic treatment phase (Week 2 up to Week 5 - visit 2 to visit 3): At week 2, all the subjects will start to apply a topical antibiotic (Neomycin/Nebacetin® ointment) for the next 3 weeks.
  * Treatment phase 2 (from week 5 up to week 13 - visit 3 up to visit 5):
  Sunscreen alone will be applied again (group 1) for a minimum of 4 weeks and up to 8 weeks, according to the Global Improvement of solar lentigines and absence of PIH.
  Interventions: Procedure: Cryotherapy (CRY-AC3® device)

INTERVENTIONS:
Drug: Tri-luma — Pre-procedure phase (From Baseline up to Week 2) treated daily for their solar lentigines with the investigational drug (Tri-Luma® cream) for 2 weeks.
  Post-procedure phase (From week 2 up to Week 13 - Visit )
  - Tri-Luma® cream treatment phase (from week 5 up to week 13 - visit 3 up to visit 5):The investigational drug (Tri-Luma® cream) will be applied again (group 1) for a minimum of 4 weeks and up to 8 weeks, according to the Global Improvement of solar lentigines and absence of PIH.
  Arms: Group 1
Procedure: Cryotherapy (CRY-AC3® device) — Procedure performed at week 2.

SUMMARY:
To evaluate safety and efficacy of Tri-Luma® cream as an adjunctive treatment to cryotherapy when used in the pre- and post-procedure phases for the treatment of solar lentigines on the back of the hands and in the prevention of post-inflammatory hyperpigmentation after cryotherapy.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of Tri-Luma® cream as an adjunctive treatment to cryotherapy when used in the pre- and post-procedure phases for the treatment of solar lentigines on the back of the hands and in the prevention of post-inflammatory hyperpigmentation after cryotherapy.

The study has 13 weeks for each subject. Five visits will take place: at Baseline, week 2, 5, 9 and 13 after the cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol;
* Female and male subjects;
* Phototype II to IV;
* Subjects aged between 40 and 65 years;
* Subjects presenting at least 5 lesions of solar lentigines at the back hands with al least 3mm of diameter
* History of post-inflammatory hyperpigmentation on body or face
* Medical history and physical examination which, based on the investigator's opinion, do not prevent the subject from taking part in the study or from making use of the products under investigation;
* Subjects of childbearing age should present a negative urine pregnancy test at baseline and should be using a highly effective contraceptive method during all study;
* Availability of the subject throughout the study;
* Subject agreeing not to undergo other cosmetic or dermatological procedures during the participation in the study;
* Subjects with sufficient schooling and knowledge to enable them to cooperate to the degree required by the protocol.

Exclusion Criteria:

* Pregnant women or women intending to become pregnant in the following 5 months after screening;
* Lactation period;
* Subjects participating in other clinical trials;
* Any prior cosmetic procedures, including fillers, or scars that may interfere with the study results;
* Subjects with neoplastic, muscular or neurological diseases;
* Subjects with inflammation or active infection in the area to be studied;
* Subjects with a history of adverse effects, such as sensitivity to the components of any of the study drug formula,
* Subjects with a history of non-adherence to medical treatment or showing unwillingness to adhere to the study protocol;
* Any condition that, in the opinion of the investigator, can compromise the evaluation of the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, MD, Principal Investigator — Brazilian Center for Studies in Dermatology

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Subjects treated daily for their solar lentigines with the triple combination (hydroquinone 4% tretinoin 0.05% fluocinolone acetonide 0.01%; Tri-Luma® cream) plus sunscreen for 2 weeks. At week 2, all the subjects had the solar lentigines treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (Week 2 up to Week 13)
  * Topical antibiotic treatment (Week 2 to Week 5): All the subjects applied a topical antibiotic (Neomycin/Nebacetin® ointment) for the following 3 weeks.
  * Second treatment phase (Week 5 to Week 13):
  Subjects of group 1 applied Tri-Luma® cream plus sunscreen again for a minimum of 4 weeks and up to 8 weeks, depending on the Global Improvement of solar lentigines score and absence of post inflammatory hyperpigmentation.
- Group 2: Subjects treated daily for their solar lentigines with sunscreen only for 2 weeks. At week 2, all the subjects had the solar lentigines treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (Week 2 up to Week 13)
  * Topical antibiotic treatment phase (Week 2 to Week 5): All the subjects applied a topical antibiotic (Neomycin/Nebacetin® ointment) for the next 3 weeks.
  * Second treatment phase (Week 5 to Week 13):
  Subjects of group 2 applied sunscreen only again for a minimum of 4 weeks and up to 8 weeks, depending on the Global Improvement of solar lentigines score and absence of post inflammatory hyperpigmentation.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 25 | 25
Completed | 23 | 22
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Subjects treated daily for their solar lentigines with the triple combination (hydroquinone 4% tretinoin 0.05% fluocinolone acetonide 0.01%; Tri-Luma® cream) plus sunscreen for 2 weeks. At week 2, all the subjects had the solar lentigines treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (Week 2 up to Week 13)
  * Topical antibiotic treatment (Week 2 to Week 5): All the subjects applied a topical antibiotic (Neomycin/Nebacetin® ointment) for the following 3 weeks.
  * Second treatment phase (Week 5 to Week 13):
  Subjects of group 1 applied Tri-Luma® cream plus sunscreen again for a minimum of 4 weeks and up to 8 weeks, depending on the Global Improvement of solar lentigines score and absence of PIH.
- Group 2: Subjects treated daily for their solar lentigines with sunscreen only for 2 weeks. At week 2, all the subjects had the solar lentigines treated by cryotherapy (CRY-AC3® device).
  Post-procedure phase (Week 2 up to Week 13)
  * Topical antibiotic treatment phase (Week 2 to Week 5): All the subjects applied a topical antibiotic (Neomycin/Nebacetin® ointment) for the next 3 weeks.
  * Second treatment phase (Week 5 to Week 13):
  Subjects of group 2 applied sunscreen only again for a minimum of 4 weeks and up to 8 weeks, depending on the Global Improvement of solar lentigines score and absence of PIH.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (4) | 56 (6) | 58 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 24 | 49
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Solar Lentigines Count
Description: Solar lentigines count up to 13 weeks
Time Frame: up to 13 weeks
Measure: Mean (Standard Deviation); unit: Number of solar lentigines
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 23 | 22
Number of solar lentigines
  Baseline | 25.7 (7.0) | 26.0 (11.0)
  Week 13 | 8.0 (6.0) | 11.0 (6.0)

2. Secondary Outcome: Change From Baseline in Melanin Levels
Description: This assessment was made using a narrowband reﬂectance spectrophotometer (Mexameter MX18®, Courage-Khazaka, Germany). The measurement is based on absorption/reflection. The probe of the Mexameter® MX 18 emits three specific light wavelengths. A receiver measures the light reflected by the skin. As the quantity of emitted light is defined, the quantity of light absorbed by the skin can be calculated. The melanin is measured by two specific wavelengths (red: 660 nm and near infrared: 880 nm) chosen to correspond to different absorption rates by the pigments.
  The quantification of melanin is presented as a value that varies from 0-999. The higher the value, the larger is the amount of melanin on the skin.
Time Frame: Baseline and up to 13 weeks
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 23 | 22
Arbitrary units
  Baseline | 297 (69) | 279 (68)
  Change at Week 13 | -95 (59) | -41 (65)

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=25) | Group 2 (N=25)
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2
Residual blisters from cryotherapy (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No